CLINICAL TRIAL: NCT07008196
Title: An Exploratory Clinical Study on Telitacicept for the Treatment of Refractory Rheumatoid Arthritis
Brief Title: Telitacicept for the Treatment of Refractory RA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese SLE Treatment And Research Group (Other)
Responsible Party: Principal Investigator, Xinping Tian, Professor of medicine, Chinese SLE Treatment And Research Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Telitacicept-RA
Record Dates: First submitted 2025-05-26; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis; refractory; Telitacicept
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — telitacicept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telitacicept treatment group (Experimental): Telitacicept added on previous treatment
  Interventions: Drug: Telitacicept

INTERVENTIONS:
Drug: Telitacicept — Telitacicept 160mg qw subcutaneous injection

SUMMARY:
This is a single-center, single-arm, open-label, prospective study on the efficacy and safety of Telitacicept in patients with refractory rheumatoid arthritis.

DETAILED DESCRIPTION:
The treatment of rheumatoid arthritis (RA) has made significant progress over the past three decades. However, approximately 20-30% of patients remain resistant to conventional synthetic disease-modifying antirheumatic drugs (csDMARDs), biologic DMARDs (bDMARDs), and targeted synthetic DMARDs (tsDMARDs), presenting a major challenge in RA management. Telitacicept is a dual-target inhibitor of B-cell activating factor (BAFF) and a proliferation-inducing ligand (APRIL). By inhibiting B cell maturation, differentiation, and antibody secretion by plasma cells, it reduces autoantibody production and the release of pro-inflammatory cytokines such as Tumor necrosis factor-α (TNF-α) and Interleukin-6 (IL-6), thereby alleviating joint inflammation. Clinically, a Phase III study of telitacicept in RA patients with inadequate response to methotrexate demonstrated a rapid onset of action within 4 weeks. At week 24, the ACR20 response rate in the 160 mg telitacicept group reached 67.4%, and at week 48, the response rate increased to 72.2%. Nearly 90% of patients exhibited no radiographic progression. In terms of safety, the incidence of adverse events with telitacicept was comparable to that of conventional therapies.

Currently, there are no clinical trials or registered studies investigating the use of telitacicept in the treatment of refractory RA. This study aims to evaluate the efficacy and safety of telitacicept in patients with refractory rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfill the classification criteria of the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR)
2. Refractory RA definition: Insufficient response to a combination of at least two adequate doses of csDMARDs followed by bDMARDs (including but not limited to tumor necrosis factor inhibitors, interleukin-6 receptor inhibitors, T-cell costimulation molecule inhibitors, B-cell targeted drugs) or tsDMARDs (including but not limited to JAK inhibitors) for 12 weeks, with stable drug dosage for at least 6 weeks
3. For patients treated with glucocorticoid therapy, they must have been on a stable dose of prednisone or prednisone equivalent ≤ 10 mg/day for at least 4 weeks before enrollment
4. For patients treated with non-steroidal anti-inflammatory drugs, they must have been on a stable dose for at least 2 weeks before screening and enrollment
5. ① Age > 18 years and < 70 years; ② Absolute neutrophil count ≥ 1.0 × 10⁹/L, platelet count ≥ 100 × 10⁹/L, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within 3 times the upper limit of normal, total bilirubin within 1.5 times the upper limit of normal, serum creatinine clearance rate > 60 ml/min; ③ Voluntarily sign the informed consent form

Exclusion Criteria:

1. Subjects with other autoimmune diseases
2. Subjects with severe and poorly controlled cardiovascular, cerebrovascular, respiratory, liver, kidney, gastrointestinal, endocrine, hematological, or neurological diseases, or laboratory abnormalities that, in the opinion of the investigator, pose unacceptable risks for participation in the study
3. Subjects with a history of malignancy (or less than 5 years since clinical remission)
4. Subjects who are pregnant or breastfeeding, or plan to become pregnant or start breastfeeding during the study period
5. Subjects who have received live virus vaccines within 4 weeks prior to enrollment in the study
6. Subjects allergic to talizumab or any excipients
7. Subjects who have participated in any other investigational drug trial within 12 weeks prior to the start of this study
8. Subjects with active hepatitis or a history of severe liver disease at screening
9. Subjects in the active phase of herpes zoster infection, or those who have experienced severe infections (requiring intravenous antibiotics or hospitalization) within 12 weeks prior to the start of the study medication
10. Subjects with other conditions deemed unsuitable for enrollment by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
ACR20 at week 12 | Week 12
  ACR20 is a comprehensive index defined as an improvement of at least 20% in both the number of tender and swollen joints, and improvement in at least three of the following five parameters by at least 20%: 1) Visual Analogue Scale (VAS) for pain, 2) patient's global assessment, 3) physician's global assessment, 4) Health Assessment Questionnaire (HAQ), and 5) acute-phase reactants (erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP)).

SECONDARY OUTCOMES:
ACR20 at week 24 | Week 24
  ACR20 is a comprehensive index defined as an improvement of at least 20% in both the number of tender and swollen joints, and improvement in at least three of the following five parameters by at least 20%: 1) Visual Analogue Scale (VAS) for pain, 2) patient's global assessment, 3) physician's global assessment, 4) Health Assessment Questionnaire (HAQ), and 5) acute-phase reactants (erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP)).
The proportion of patients achieving DAS28 remission or low disease activity at week 12 and week 24 | Week 12 and 24
  DAS28 evaluates RA severity by quantifying joint inflammation and systemic markers of disease activity.
The proportion of patients achieving SDAI remission or low disease activity at week 12 and week 24 | Week 12 and 24
  Simplified Disease Activity Index (SDAI) is calculated by summing five parameters: Tender Joint Count (TJC28): Number of tender joints out of 28 assessed joints. Swollen Joint Count (SJC28): Number of swollen joints out of 28 assessed joints. Patient Global Assessment (PGA): Patient's self-rated health status on a 0-10 scale (0 = best, 10 = worst). Physician Global Assessment (MDGA): Physician's evaluation of disease activity on a 0-10 scale (0 = best, 10 = worst). C-reactive Protein (CRP): Laboratory value measured in mg/L.
ACR50 at week 12 and 24 | Week 12 and 24
  ACR50 is a comprehensive index defined as an improvement of at least 50% in both the number of tender and swollen joints, and improvement in at least three of the following five parameters by at least 50%: 1) Visual Analogue Scale (VAS) for pain, 2) patient's global assessment, 3) physician's global assessment, 4) Health Assessment Questionnaire (HAQ), and 5) acute-phase reactants (erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP)).
ACR70 at week 12 and 24 | Week 12 and 24
  ACR70 is a comprehensive index defined as an improvement of at least 70% in both the number of tender and swollen joints, and improvement in at least three of the following five parameters by at least 70%: 1) Visual Analogue Scale (VAS) for pain, 2) patient's global assessment, 3) physician's global assessment, 4) Health Assessment Questionnaire (HAQ), and 5) acute-phase reactants (erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP)).
The proportion of patients achieving CDAI remission or low disease activity at week 12 and week 24 | Week 12 and 24
  Clinical Disease Activity Index (CDAI) is a composite score used to assess disease activity in rheumatoid arthritis (RA). It calculates disease severity through the following parameters: Tender Joint Count (TJC28): Number of tender joints out of 28 assessed joints. Swollen Joint Count (SJC28): Number of swollen joints out of 28 assessed joints. Patient Global Assessment (PGA): Patient's self-rated health status on a 0-10 scale (0 = best, 10 = worst). Physician Global Assessment (MDGA): Physician's evaluation of disease activity on a 0-10 scale (0 = best, 10 = worst).
Change in glucocorticoid dosage | week 24
  Change in glucocorticoid dosage at week 24 of treatment compared to baseline
Adverse events | during the study period and within 4 weeks after study completion
  The incidence of all adverse events, serious adverse events, and the probability of drug discontinuation due to adverse events or serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xinping Tian, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No